CLINICAL TRIAL: NCT00293137
Title: Nitric Oxide-Derived Oxidants and Regional Endothelial and Diastolic Dysfunction in Dilated Cardiomyopathy
Brief Title: NORDIC: Nitric Oxide-Derived Oxidants and Regional Endothelial and Diastolic Dysfunction in Dilated Cardiomyopathy
Acronym: NORDIC
Status: Terminated | Type: Observational
Why Stopped: safety concerns regarding use of rosiglitazone
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Anne Kanderian, MD, Cleveland CLinic
Other Study IDs: NORDIC
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Chronic Systolic Heart Failure (Dilated Cardiomyopathy)
Keywords: Chronic systolic heart failure; Heart Failure
MeSH Terms: conditions — Cardiomyopathy, Dilated; Heart Failure

GROUPS / COHORTS (1):
- 1: Patients enrolled into the trial must have left ventricular ejection fraction of <40% by echocardiogram within 6 months of enrollment

SUMMARY:
The principal aim is to investigate the safety and efficacy of rosiglitazone in patients with chronic systolic heart (Dilated cardiomyopathy). We hypothesize that in patients with heart failure, rosiglitazone is safe, and can reduce nitric oxide (NO) derived oxidative stress (in particular, nitrotyrosine) thereby improving endothelial dysfunction, left ventricular performance, and metabolic parameters.

DETAILED DESCRIPTION:
The study will be a single center, double-blind, prospective placebo controlled trial of 60 non-diabetic heart failure patients. Prior to administration of study medication, a medical history, physician exam, blood draw, laser Doppler imaging (Periscan system), venous occlusion strain gauge plethysmography, metabolic exercise stress test and 2D and 3D echocardiograms will be performed. Patients will then be randomized to receive rosiglitazone 2mg/day oral versus placebo with up-titration to 4mg/day oral versus placebo at 3 months. Each study arm will have 30 patients who will participate for 6 months. Follow up assessments will be completed at 6 weeks, 3 months and 6 months post randomization.

ELIGIBILITY:
Inclusion Criteria:

Patients enrolled into the trial must meet all of the following criteria:

1. Chronic, stable, euvolemic, heart failure optimally treated for at least 3 months with stable doses of ACE inhibitors or angiotensin-receptor blockers and beta-blockers
2. Mild-to-moderate signs and/or symptoms of heart failure (NYHA functional Class I-II)
3. Left ventricular ejection fraction of <40% by echocardiogram within 6 months of randomization or enrollment

Exclusion Criteria:

Patients meeting one or more of the following criteria are not eligible for randomization into the trial:

1. Known or confirmed newly-diagnosed diabetes mellitus (2004 ADA criteria)
2. Major cardiovascular event (myocardial infarction, unstable angina, stroke, transient ischemic attack, pulmonary embolism), or major surgery <1 month of enrollment
3. Hospitalization or emergency room visits for heart failure exacerbation, or use of inotropic agents < 1 month
4. NYHA class III or IV
5. Current treatment with thiazolidinediones
6. Allergy to rosiglitazone, or liver insufficiency (ALT > 2.5x upper limits of normal)
7. Heart failure due to congenital heart disease, primary valvular disease, hypertrophic cardiomyopathy, or heart failure caused by known cardiotoxic agents (e.g. adriamycin)
8. End-stage renal failure on renal replacement therapy (dialysis)
9. Life expectancy, or expected cardiac transplantation within 12 months of enrollment
10. Women who are pregnant, or who are planning on becoming pregnant or are lactating. Women of childbearing potential must have a negative serum pregnancy test within 48 hours prior to the time of randomization and must use contraceptive agents
11. Unable or unwilling to consent to all components of the protocol. Patients unwilling to undergo 6-month follow-up should not be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: see inclusion/exclusion
Enrollment: 60 (Estimated)
Dates: Start 2006-02; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint • Comparison of NO-derived oxidants, systemic ADMA, skin blood flow, forearm blood flow and exhaled NO. • Correlation of NO-derived oxidants, systemic ADMA, skin blood flow, forearm blood flow and exhaled NO to functional capacity | 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Wilson H Tang, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States